CLINICAL TRIAL: NCT04629261
Title: Effects of the Mexico City´s ECOBICI Program on Health Indicators and Physical Activity Levels
Brief Title: Effects of Bicycle-sharing Program on Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Catalina Medina, MSc, PhD, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECOBICI and Health
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity
Keywords: Shared bicycle systems; Physical activity; Body mass index; Blood pressure; Eating habits; Commuting cycling
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial: 2 intervention groups and 1 control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Users with no incentive (Experimental): Participants who are interested on get involved into the ECOBICI program, and who randomly will not receive a discount fee for enrollment.
  Interventions: Behavioral: Use of ECOBICI (public bicycle sharing program)
- Users with incentive (Experimental): Participants who are interested on get involved into the ECOBICI program, and who randomly will do receive a discount fee for enrollment.
  Interventions: Behavioral: Use of ECOBICI (public bicycle sharing program)
- Non-users (No Intervention): Participants with an age range similar to the intervention groups, who work or lives nearby ECOBICI's bicycle station, that are not enrolled in the ECOBICI program or in a health related program (ex. reducing weight).

INTERVENTIONS:
Behavioral: Use of ECOBICI (public bicycle sharing program) — Use of ECOBICI program with and without incentive.
  Arms: Users with incentive; Users with no incentive

SUMMARY:
To evaluate the effect of the ECOBICI program in Mexico City on health indicators, activity levels, mental health, and quality of life and diet after 3 months of follow-up.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) such as obesity and type 2 diabetes mellitus (DM2) are one of the main causes of death in the world and in Mexico. According to the 2016 National Health and Nutrition Survey (ENSANUT), 9.4% has previously diagnosed diabetes and the prevalence of overweight and obesity is 71.2% in adults. Among the main risk factors for the development of these diseases are an unbalanced diet, physical inactivity and sedentarism.

According to the World Health Organization (WHO), accumulating at least 150 minutes/week of moderate-vigorous physical activity either during occupational, home, leisure time and transportation for at least 10 continuous minutes could result multiple benefits, such as the reduction of seven types of NCDs including DM2 and obesity. It has been observed that cycling, compared to other activities during leisure time, appears to be an efficient form of daily exercise and feasible to increase physical activity levels even in the most physically inactive individuals.

According to a cross-sectional study in 14 countries including the United States, it was observed that adults who commuted by bicycle had a lower risk of DM2 and obesity. Additionally, results from randomized controlled studies have shown that cycling may help reducing body fat and increase maximal oxygen consumption. However, some factors, such as the lack of attractive bike paths and the lack of safe spaces, may reduce this pattern.

The shared bicycle program has been implemented in more than 30 countries including Mexico. Among the main objectives of this program - in addition to integrating the bicycle as a form of active transportation - includes the design of a new infrastructure to offer safety and comfort to cyclists. This type of program has been evaluated in different countries. Results show that the combination of interventions, that is, the construction of bicycle facilities and the shared bicycle programs increased trips in Barcelona and Paris. In Barcelona, it was observed that this program increased the quality of life and decreased air and noise pollution. In Montreal, this program was found to attract young people and people within the highest socioeconomic status. In Valencia, Spain, it was reported that the bicycle system increased energy expenditure by 257 METs / min / week and helped reducing 2kg. of body weight in a school year. In Japan, pedaling for 30 minutes to work was found to have an effect on mental health. Finally, in the United States, it was observed that those who use active transportation to go to work have a lower probability of obesity, elevated triglyceride levels, diastolic blood pressure, and fasting glucose.

The ECOBICI program is a shared bicycle system within Mexico City. Since 2010, this program has been managed by the Ministry of Environment and the Ministry of Mobility, initially operating with 1,200 bicycles and 84 bicycle stations around Mexico City. It currently belongs to the Comprehensive Mobility Program 2018-2024, aiming at the accessibility of the population in the use of bicycles, promoting their use as an air pollution free transport. This program has been awarded within the urban public transport area, for improving air quality and for seeking a change in society.

Authorities of the ECOBICI program conducted a users' survey in 2014, this included questions related to the program and health aspects of the users. It was observed that 36% of those surveyed perceived an improvement in their physical condition, 15% reported having an improvement in their health and 8% reported having lost weight, however, to date there are few prospective studies that report the effect of the use of public bicycles on the levels of physical activity and health indicators.

Procedure The project is divided into two phases: phase 1 - initial evaluations and phase 2 - follow-up. Through social media (twitter and Facebook) adults interested on getting involved in the ECOBICI program and adults who are not involved in the program or physical activities aimed to improve their health will be invited to participate. All individuals interested on participating in this study will received an email indicating a day and time for a zoom meeting. The investigators will perform two zoom meetings, one for the intervention group and another for the control group. Within the intervention group meeting the investigators will explain them the study, benefits and risks to participate and the investigators will randomly allocate adults in intervention group 1 (free annual program fee) and intervention group 2 (annual program fee paid by participants). Within the control group meeting the investigators will explain them the study, benefits and risks to participate.

PHASE 1 (month 0). All adults who agree to participate must read and sign the consent letter before getting involved into the study. Then, the investigators will ask participants to answer a 20-minutes long questionnaire and will perform anthropometric and blood pressure measurements. All participants will be evaluated in the ECOBICI module considering COVID-19 hygiene guidelines. At the end of this phase, adults will be invited to participate in PHASE 2 of the study. If agree to participate, the investigator will ask for their cell phone number or home phone number to be contacted later.

PHASE 2 (months 1.5 and 3). The investigators will ask them if we could monitor their bicycle trajectories using the data from the Ministry of Mobility. In addition, the investigators will ask adults to use the STRAVA app (GPS app that monitors bike paths) every time they ride the bike. A manual will be send by email within instructions on how to download the application and how to use it. In addition, they will be instructed to send us by email the bike trajectories stored in the STRAVA application.

During month 1.5, the investigators will call them to conduct another survey focused on physical activity levels, diet, mental health, and health indicators (same survey that was conducted in month 0).

In month 3, the investigators will quote the patients in the ECOBICI module, within this visit a final questionnaire and anthropometric and blood pressure measurements will carry out.

All people who agree to participate in the TWO PHASES of the study will receive a voucher for $ 250 pesos ($1.25 USD).

ELIGIBILITY:
Inclusion criteria for intervention groups:

* Interested on getting involved in the ECOBICI program.

Exclusion criteria for intervention groups:

* Present any physical or mental condition that inhibits cycling.

Elimination criteria for intervention groups:

* Have participated only in phase one.

Inclusion Criteria for control group:

* Participants located near by program bike-stations.
* Age range similar to the intervention group.
* Not enrolled in the ECOBICI program.
* Not enrolled in an exercise program or do physical activity aimed to improve health.

Elimination criteria for control group:

* Have participated only in phase one.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity not related to the bicycle sharing program | up to 1.5 months.
  Assessed by questionnaire and expressed in minutes per week
Physical activity not related to the bicycle sharing program | up to 3 months.
  Assessed by questionnaire and expressed in minutes per week
Physical activity of bicycle sharing program | up to 1.5 months.
  Assessed by questionnaire and daily monitoring of the users' trips through automatic system records done at bike-stations of the program and by a mobile GPS application. Expressed in kilometers per trip per day and time in minutes per trip per date.
Physical activity of bicycle sharing program | up to 3 months.
  Assessed by questionnaire and daily monitoring of the users' trips through automatic system records done at bike-stations of the program and by a mobile GPS application. Expressed in kilometers per trip per day and time in minutes per trip per date.
Changes in body mass index | up to 3 months.
  Assessed by direct measurements done by trained staff and expressed in kg/m^2. Classified according to the following criteria: low weight if it´s <18.5 kg/m^2, normal if it goes from 18.5 to 24.9 kg /m^2 , overweight if it goes from 25 to 29.9 kg/m^2 or obese if it´s >30 kg/m^2.
Changes in blood pressure | up to 3 months.
  Assessed by direct measurements done by trained staff and expressed in mmHg. Classified with each participant's result according to the following criteria: normotensive if the systolic blood pressure (SBP) is <140 mmHg and diastolic blood pressure (DBP) <90 mmHg or hypertensive if the SBP is ≥140 mmHg or DBP ≥90 mmHg.
Changes in waist circumference | up to 3 months.
  Assessed by direct measurements done by trained staff and expressed in cm. Classified as high if > 92 centimeters (cm) for men or > 80 cm for women.
Changes in hip circumference | up to 3 months.
  Assessed by direct measurements done by trained staff and expressed in cm.
Changes in mental health status | up to 1.5 months.
  Assessed by questionnaire. Expressed by a general score. Depression if ≥9 for adults and ≥5 for older adults.
Changes in mental health status | up to 3 months.
  Assessed by questionnaire. Expressed by a general score. Depression if ≥9 for adults and ≥5 for older adults.
Changes in physical health | up to 1.5 months.
  Assessed by questionnaire. Expressed by a percentage.
Changes in physical health. | up to 3 months.
  Assessed by questionnaire. Expressed by a percentage.
Changes in general health status. | up to 1.5 months.
  Assessed by questionnaire. Expressed by a percentage.
Changes in general health status. | up to 3 months.
  Assessed by questionnaire. Expressed by a percentage.
Changes quality of life | up to 3 months.
  Assessed by questionnaire. Expressed by a percentage. Good and bad

SECONDARY OUTCOMES:
Changes in dietary patterns | up to 1.5 months.
  Assessed by a a semi-quantitative food frequency questionnaire. Expressed by a percentage.
Changes in dietary patterns | up to 3 months.
  Assessed by a a semi-quantitative food frequency questionnaire. Expressed by a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Catalina Medina, Ph.D., Principal Investigator — Instituto Nacional de Salud Pública

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barquera S, Pedroza-Tobias A, Medina C. Cardiovascular diseases in mega-countries: the challenges of the nutrition, physical activity and epidemiologic transitions, and the double burden of disease. Curr Opin Lipidol. 2016 Aug;27(4):329-44. doi: 10.1097/MOL.0000000000000320. PMID 27389629
- [Background] Barquera S, Campos-Nonato I, Hernandez-Barrera L, Pedroza A, Rivera-Dommarco JA. [Prevalence of obesity in Mexican adults 2000-2012]. Salud Publica Mex. 2013;55 Suppl 2:S151-60. Spanish. PMID 24626691
- [Background] GBD 2013 Risk Factors Collaborators; Forouzanfar MH, Alexander L, Anderson HR, Bachman VF, Biryukov S, Brauer M, Burnett R, Casey D, Coates MM, Cohen A, Delwiche K, Estep K, Frostad JJ, Astha KC, Kyu HH, Moradi-Lakeh M, Ng M, Slepak EL, Thomas BA, Wagner J, Aasvang GM, Abbafati C, Abbasoglu Ozgoren A, Abd-Allah F, Abera SF, Aboyans V, Abraham B, Abraham JP, Abubakar I, Abu-Rmeileh NM, Aburto TC, Achoki T, Adelekan A, Adofo K, Adou AK, Adsuar JC, Afshin A, Agardh EE, Al Khabouri MJ, Al Lami FH, Alam SS, Alasfoor D, Albittar MI, Alegretti MA, Aleman AV, Alemu ZA, Alfonso-Cristancho R, Alhabib S, Ali R, Ali MK, Alla F, Allebeck P, Allen PJ, Alsharif U, Alvarez E, Alvis-Guzman N, Amankwaa AA, Amare AT, Ameh EA, Ameli O, Amini H, Ammar W, Anderson BO, Antonio CA, Anwari P, Argeseanu Cunningham S, Arnlov J, Arsenijevic VS, Artaman A, Asghar RJ, Assadi R, Atkins LS, Atkinson C, Avila MA, Awuah B, Badawi A, Bahit MC, Bakfalouni T, Balakrishnan K, Balalla S, Balu RK, Banerjee A, Barber RM, Barker-Collo SL, Barquera S, Barregard L, Barrero LH, Barrientos-Gutierrez T, Basto-Abreu AC, Basu A, Basu S, Basulaiman MO, Batis Ruvalcaba C, Beardsley J, Bedi N, Bekele T, Bell ML, Benjet C, Bennett DA, Benzian H, Bernabe E, Beyene TJ, Bhala N, Bhalla A, Bhutta ZA, Bikbov B, Bin Abdulhak AA, Blore JD, Blyth FM, Bohensky MA, Bora Basara B, Borges G, Bornstein NM, Bose D, Boufous S, Bourne RR, Brainin M, Brazinova A, Breitborde NJ, Brenner H, Briggs AD, Broday DM, Brooks PM, Bruce NG, Brugha TS, Brunekreef B, Buchbinder R, Bui LN, Bukhman G, Bulloch AG, Burch M, Burney PG, Campos-Nonato IR, Campuzano JC, Cantoral AJ, Caravanos J, Cardenas R, Cardis E, Carpenter DO, Caso V, Castaneda-Orjuela CA, Castro RE, Catala-Lopez F, Cavalleri F, Cavlin A, Chadha VK, Chang JC, Charlson FJ, Chen H, Chen W, Chen Z, Chiang PP, Chimed-Ochir O, Chowdhury R, Christophi CA, Chuang TW, Chugh SS, Cirillo M, Classen TK, Colistro V, Colomar M, Colquhoun SM, Contreras AG, Cooper C, Cooperrider K, Cooper LT, Coresh J, Courville KJ, Criqui MH, Cuevas-Nasu L, Damsere-Derry J, Danawi H, Dandona L, Dandona R, Dargan PI, Davis A, Davitoiu DV, Dayama A, de Castro EF, De la Cruz-Gongora V, De Leo D, de Lima G, Degenhardt L, del Pozo-Cruz B, Dellavalle RP, Deribe K, Derrett S, Des Jarlais DC, Dessalegn M, deVeber GA, Devries KM, Dharmaratne SD, Dherani MK, Dicker D, Ding EL, Dokova K, Dorsey ER, Driscoll TR, Duan L, Durrani AM, Ebel BE, Ellenbogen RG, Elshrek YM, Endres M, Ermakov SP, Erskine HE, Eshrati B, Esteghamati A, Fahimi S, Faraon EJ, Farzadfar F, Fay DF, Feigin VL, Feigl AB, Fereshtehnejad SM, Ferrari AJ, Ferri CP, Flaxman AD, Fleming TD, Foigt N, Foreman KJ, Paleo UF, Franklin RC, Gabbe B, Gaffikin L, Gakidou E, Gamkrelidze A, Gankpe FG, Gansevoort RT, Garcia-Guerra FA, Gasana E, Geleijnse JM, Gessner BD, Gething P, Gibney KB, Gillum RF, Ginawi IA, Giroud M, Giussani G, Goenka S, Goginashvili K, Gomez Dantes H, Gona P, Gonzalez de Cosio T, Gonzalez-Castell D, Gotay CC, Goto A, Gouda HN, Guerrant RL, Gugnani HC, Guillemin F, Gunnell D, Gupta R, Gupta R, Gutierrez RA, Hafezi-Nejad N, Hagan H, Hagstromer M, Halasa YA, Hamadeh RR, Hammami M, Hankey GJ, Hao Y, Harb HL, Haregu TN, Haro JM, Havmoeller R, Hay SI, Hedayati MT, Heredia-Pi IB, Hernandez L, Heuton KR, Heydarpour P, Hijar M, Hoek HW, Hoffman HJ, Hornberger JC, Hosgood HD, Hoy DG, Hsairi M, Hu G, Hu H, Huang C, Huang JJ, Hubbell BJ, Huiart L, Husseini A, Iannarone ML, Iburg KM, Idrisov BT, Ikeda N, Innos K, Inoue M, Islami F, Ismayilova S, Jacobsen KH, Jansen HA, Jarvis DL, Jassal SK, Jauregui A, Jayaraman S, Jeemon P, Jensen PN, Jha V, Jiang F, Jiang G, Jiang Y, Jonas JB, Juel K, Kan H, Kany Roseline SS, Karam NE, Karch A, Karema CK, Karthikeyan G, Kaul A, Kawakami N, Kazi DS, Kemp AH, Kengne AP, Keren A, Khader YS, Khalifa SE, Khan EA, Khang YH, Khatibzadeh S, Khonelidze I, Kieling C, Kim D, Kim S, Kim Y, Kimokoti RW, Kinfu Y, Kinge JM, Kissela BM, Kivipelto M, Knibbs LD, Knudsen AK, Kokubo Y, Kose MR, Kosen S, Kraemer A, Kravchenko M, Krishnaswami S, Kromhout H, Ku T, Kuate Defo B, Kucuk Bicer B, Kuipers EJ, Kulkarni C, Kulkarni VS, Kumar GA, Kwan GF, Lai T, Lakshmana Balaji A, Lalloo R, Lallukka T, Lam H, Lan Q, Lansingh VC, Larson HJ, Larsson A, Laryea DO, Lavados PM, Lawrynowicz AE, Leasher JL, Lee JT, Leigh J, Leung R, Levi M, Li Y, Li Y, Liang J, Liang X, Lim SS, Lindsay MP, Lipshultz SE, Liu S, Liu Y, Lloyd BK, Logroscino G, London SJ, Lopez N, Lortet-Tieulent J, Lotufo PA, Lozano R, Lunevicius R, Ma J, Ma S, Machado VM, MacIntyre MF, Magis-Rodriguez C, Mahdi AA, Majdan M, Malekzadeh R, Mangalam S, Mapoma CC, Marape M, Marcenes W, Margolis DJ, Margono C, Marks GB, Martin RV, Marzan MB, Mashal MT, Masiye F, Mason-Jones AJ, Matsushita K, Matzopoulos R, Mayosi BM, Mazorodze TT, McKay AC, McKee M, McLain A, Meaney PA, Medina C, Mehndiratta MM, Mejia-Rodriguez F, Mekonnen W, Melaku YA, Meltzer M, Memish ZA, Mendoza W, Mensah GA, Meretoja A, Mhimbira FA, Micha R, Miller TR, Mills EJ, Misganaw A, Mishra S, Mohamed Ibrahim N, Mohammad KA, Mokdad AH, Mola GL, Monasta L, Montanez Hernandez JC, Montico M, Moore AR, Morawska L, Mori R, Moschandreas J, Moturi WN, Mozaffarian D, Mueller UO, Mukaigawara M, Mullany EC, Murthy KS, Naghavi M, Nahas Z, Naheed A, Naidoo KS, Naldi L, Nand D, Nangia V, Narayan KM, Nash D, Neal B, Nejjari C, Neupane SP, Newton CR, Ngalesoni FN, Ngirabega Jde D, Nguyen G, Nguyen NT, Nieuwenhuijsen MJ, Nisar MI, Nogueira JR, Nolla JM, Nolte S, Norheim OF, Norman RE, Norrving B, Nyakarahuka L, Oh IH, Ohkubo T, Olusanya BO, Omer SB, Opio JN, Orozco R, Pagcatipunan RS Jr, Pain AW, Pandian JD, Panelo CI, Papachristou C, Park EK, Parry CD, Paternina Caicedo AJ, Patten SB, Paul VK, Pavlin BI, Pearce N, Pedraza LS, Pedroza A, Pejin Stokic L, Pekericli A, Pereira DM, Perez-Padilla R, Perez-Ruiz F, Perico N, Perry SA, Pervaiz A, Pesudovs K, Peterson CB, Petzold M, Phillips MR, Phua HP, Plass D, Poenaru D, Polanczyk GV, Polinder S, Pond CD, Pope CA, Pope D, Popova S, Pourmalek F, Powles J, Prabhakaran D, Prasad NM, Qato DM, Quezada AD, Quistberg DA, Racape L, Rafay A, Rahimi K, Rahimi-Movaghar V, Rahman SU, Raju M, Rakovac I, Rana SM, Rao M, Razavi H, Reddy KS, Refaat AH, Rehm J, Remuzzi G, Ribeiro AL, Riccio PM, Richardson L, Riederer A, Robinson M, Roca A, Rodriguez A, Rojas-Rueda D, Romieu I, Ronfani L, Room R, Roy N, Ruhago GM, Rushton L, Sabin N, Sacco RL, Saha S, Sahathevan R, Sahraian MA, Salomon JA, Salvo D, Sampson UK, Sanabria JR, Sanchez LM, Sanchez-Pimienta TG, Sanchez-Riera L, Sandar L, Santos IS, Sapkota A, Satpathy M, Saunders JE, Sawhney M, Saylan MI, Scarborough P, Schmidt JC, Schneider IJ, Schottker B, Schwebel DC, Scott JG, Seedat S, Sepanlou SG, Serdar B, Servan-Mori EE, Shaddick G, Shahraz S, Levy TS, Shangguan S, She J, Sheikhbahaei S, Shibuya K, Shin HH, Shinohara Y, Shiri R, Shishani K, Shiue I, Sigfusdottir ID, Silberberg DH, Simard EP, Sindi S, Singh A, Singh GM, Singh JA, Skirbekk V, Sliwa K, Soljak M, Soneji S, Soreide K, Soshnikov S, Sposato LA, Sreeramareddy CT, Stapelberg NJ, Stathopoulou V, Steckling N, Stein DJ, Stein MB, Stephens N, Stockl H, Straif K, Stroumpoulis K, Sturua L, Sunguya BF, Swaminathan S, Swaroop M, Sykes BL, Tabb KM, Takahashi K, Talongwa RT, Tandon N, Tanne D, Tanner M, Tavakkoli M, Te Ao BJ, Teixeira CM, Tellez Rojo MM, Terkawi AS, Texcalac-Sangrador JL, Thackway SV, Thomson B, Thorne-Lyman AL, Thrift AG, Thurston GD, Tillmann T, Tobollik M, Tonelli M, Topouzis F, Towbin JA, Toyoshima H, Traebert J, Tran BX, Trasande L, Trillini M, Trujillo U, Dimbuene ZT, Tsilimbaris M, Tuzcu EM, Uchendu US, Ukwaja KN, Uzun SB, van de Vijver S, Van Dingenen R, van Gool CH, van Os J, Varakin YY, Vasankari TJ, Vasconcelos AM, Vavilala MS, Veerman LJ, Velasquez-Melendez G, Venketasubramanian N, Vijayakumar L, Villalpando S, Violante FS, Vlassov VV, Vollset SE, Wagner GR, Waller SG, Wallin MT, Wan X, Wang H, Wang J, Wang L, Wang W, Wang Y, Warouw TS, Watts CH, Weichenthal S, Weiderpass E, Weintraub RG, Werdecker A, Wessells KR, Westerman R, Whiteford HA, Wilkinson JD, Williams HC, Williams TN, Woldeyohannes SM, Wolfe CD, Wong JQ, Woolf AD, Wright JL, Wurtz B, Xu G, Yan LL, Yang G, Yano Y, Ye P, Yenesew M, Yentur GK, Yip P, Yonemoto N, Yoon SJ, Younis MZ, Younoussi Z, Yu C, Zaki ME, Zhao Y, Zheng Y, Zhou M, Zhu J, Zhu S, Zou X, Zunt JR, Lopez AD, Vos T, Murray CJ. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Dec 5;386(10010):2287-323. doi: 10.1016/S0140-6736(15)00128-2. Epub 2015 Sep 11. PMID 26364544
- [Background] Warburton DE, Charlesworth S, Ivey A, Nettlefold L, Bredin SS. A systematic review of the evidence for Canada's Physical Activity Guidelines for Adults. Int J Behav Nutr Phys Act. 2010 May 11;7:39. doi: 10.1186/1479-5868-7-39. PMID 20459783
- [Background] Moller NC, Ostergaard L, Gade JR, Nielsen JL, Andersen LB. The effect on cardiorespiratory fitness after an 8-week period of commuter cycling--a randomized controlled study in adults. Prev Med. 2011 Sep;53(3):172-7. doi: 10.1016/j.ypmed.2011.06.007. Epub 2011 Jun 25. PMID 21708185
- [Background] Pucher J, Buehler R, Bassett DR, Dannenberg AL. Walking and cycling to health: a comparative analysis of city, state, and international data. Am J Public Health. 2010 Oct;100(10):1986-92. doi: 10.2105/AJPH.2009.189324. Epub 2010 Aug 19. PMID 20724675
- [Background] Molina-Garcia J, Castillo I, Sallis JF. Psychosocial and environmental correlates of active commuting for university students. Prev Med. 2010 Aug;51(2):136-8. doi: 10.1016/j.ypmed.2010.05.009. Epub 2010 May 25. PMID 20510271
- [Background] Pucher J, Dill J, Handy S. Infrastructure, programs, and policies to increase bicycling: an international review. Prev Med. 2010 Jan;50 Suppl 1:S106-25. doi: 10.1016/j.ypmed.2009.07.028. Epub 2009 Sep 16. PMID 19765610
- [Background] Fuller D, Gauvin L, Kestens Y, Daniel M, Fournier M, Morency P, Drouin L. Use of a new public bicycle share program in Montreal, Canada. Am J Prev Med. 2011 Jul;41(1):80-3. doi: 10.1016/j.amepre.2011.03.002. PMID 21665067
- [Background] Molina-Garcia J, Castillo I, Queralt A, Sallis JF. Bicycling to university: evaluation of a bicycle-sharing program in Spain. Health Promot Int. 2015 Jun;30(2):350-8. doi: 10.1093/heapro/dat045. Epub 2013 Jun 28. PMID 23813668
- [Background] Ohta M, Mizoue T, Mishima N, Ikeda M. Effect of the physical activities in leisure time and commuting to work on mental health. J Occup Health. 2007 Jan;49(1):46-52. doi: 10.1539/joh.49.46. PMID 17314466
- [Background] Deramond H, Depriester C, Galibert P, Le Gars D. Percutaneous vertebroplasty with polymethylmethacrylate. Technique, indications, and results. Radiol Clin North Am. 1998 May;36(3):533-46. doi: 10.1016/s0033-8389(05)70042-7. PMID 9597071
- [Background] GBD 2015 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1659-1724. doi: 10.1016/S0140-6736(16)31679-8. PMID 27733284
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Haseler C, Crooke R, Haseler T. Promoting physical activity to patients. BMJ. 2019 Sep 17;366:l5230. doi: 10.1136/bmj.l5230. No abstract available. PMID 31530549
- [Background] Ferrari de Lima D, Anguera Lima L, do Carmo Luiz O. Daily physical activity of Brazilian carriers of arterial hypertension: a transversal analysis. Colomb Med (Cali). 2017 Jun 30;48(2):82-87. PMID 28883668
- [Background] Wen LM, Rissel C. Inverse associations between cycling to work, public transport, and overweight and obesity: findings from a population based study in Australia. Prev Med. 2008 Jan;46(1):29-32. doi: 10.1016/j.ypmed.2007.08.009. Epub 2007 Aug 23. PMID 17904210
- [Background] Sarmiento OL, Diaz Del Castillo A, Triana CA, Acevedo MJ, Gonzalez SA, Pratt M. Reclaiming the streets for people: Insights from Ciclovias Recreativas in Latin America. Prev Med. 2017 Oct;103S:S34-S40. doi: 10.1016/j.ypmed.2016.07.028. Epub 2016 Aug 3. PMID 27497659
- [Background] Atherosclerosis, Hypertension, and Obesity in the Young Committee of the American Heart Association Council on Cardiovascular Disease in the Young; Alpert B, McCrindle B, Daniels S, Dennison B, Hayman L, Jacobson M, Mahoney L, Rocchini A, Steinberger J, Urbina E, Williams R. Recommendations for blood pressure measurement in human and experimental animals; part 1: blood pressure measurement in humans. Hypertension. 2006 Jul;48(1):e3; author reply e5. doi: 10.1161/01.HYP.0000229661.06235.08. Epub 2006 Jun 12. No abstract available. PMID 16769991
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- See also: Recomendaciones mundiales sobre la actividad física para la salud. Organización Mundial de la Salud. 2010. — http://whqlibdoc.who.int/publications/2010/9789243599977_spa.pdf
- See also: Delgado Peralta M. Enseñanzas del Sistema Ecobici para la implementación de Sistemas de Bicicleta Pública en México 2016 — http://library.fes.de/pdf-files/bueros/mexiko/13013.pdf
- See also: Jefatura del Gobierno. Gaceta Oficial Distrito Federal. Administración Pública del Distrito Federal 2014. — http://www.ordenjuridico.gob.mx/Documentos/Estatal/Distrito%20Federal/wo99436.pdf
- See also: Estadísticas Ecobici. SEDEMA. — https://www.ecobici.cdmx.gob.mx/es/estadisticas
- See also: Díaz R, Rojas F. Mujeres y ciclismo urbano. Promoviendo políticas inclusivas de movilidad en América Latina. 2017 — https://publications.iadb.org/publications/spanish/document/Mujeres-y-ciclismo-urbano-Promoviendo-pol%C3%ADticas-inclusivas-de-movilidad-en-Am%C3%A9rica-Latina.pdf
- See also: Naciones Unidas. Informe de los objetivos de desarrollo sostenible 2018. — http://unstats.un.org/sdgs/files/report/2018/TheSustainableDevelopmentGoalsReport2018-ES.pdf